CLINICAL TRIAL: NCT07364357
Title: An Open-label Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of CREPT-618 in Patients With Locally Advanced Hepatocellular Carcinoma
Brief Title: A Phase I Study of CREPT-618 in Locally Advanced HCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY-618-IIT01
Record Dates: First submitted 2025-09-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CREPT-618 (Experimental): The study employs a 3+3 dose escalation design for dose titration, consisting of three primary dose groups: low dose(sentinel dose), medium dose, and high dose.Starting with the sentinel dose, one sentinel patient will be enrolled in the low-dose group and observed for up to 28 days. If no dose-limiting toxicity (DLT) occurs in the sentinel patient, enrollment will proceed. To ensure the trial can escalate to the anticipated effective dose, if no DLTs are observed in the low-, medium-, or high-dose groups, and no changes are observed in objective response rate or liver function indicators, the dose may be adjusted to a new dose.
  Interventions: Genetic: gene therapy

INTERVENTIONS:
Genetic: gene therapy — Using small nucleic acid drug to targeting CREPT

SUMMARY:
This is a single-center, open-label, dose-escalation Phase I clinical study designed to evaluate the safety (incidence of adverse events), maximum tolerated dose (MTD), optimal biological dose (OBD), and recommended Phase II dose (RP2D) of CREPT-618 in adult patients aged 18-75 with locally advanced hepatocellular carcinoma who have failed standard treatment.

The study adopts a 3+3 dose escalation design for dose climbing, primarily consisting of three dose groups: low dose, medium dose, and high dose. Patient enrollment and dose escalation in each group will be based on safety evaluation results. Pharmacokinetic parameters and preliminary efficacy indicators will also be assessed.

DETAILED DESCRIPTION:
This is a single-center, open-label, dose-escalation Phase I clinical study designed to evaluate the safety (incidence of adverse events), maximum tolerated dose (MTD), optimal biological dose (OBD), and recommended Phase II dose (RP2D) of CREPT-618 in adult patients aged 18-75 with locally advanced hepatocellular carcinoma who have failed standard treatment.

The study employs a 3+3 dose escalation design for dose titration, consisting of three primary dose groups: low dose, medium dose, and high dose. Patient enrollment and dose escalation in each cohort will be based on safety evaluation results. Pharmacokinetic parameters and preliminary efficacy indicators will also be assessed.

The study design includes three dose groups, with a total of 7-13 patients. The dose groups are divided into low dose (sentinel dose, 0.5 mg/kg), medium dose (1.5 mg/kg), and high dose (4.5 mg/kg). The low-dose group (sentinel) will enroll 1 patient; the medium-dose group, 3-6 patients; and the high-dose group, 3-6 patients. Each patient will receive single or multiple subcutaneous injections of CREPT-618 administered once every two weeks. Assessment timepoints include safety evaluations, pharmacokinetic (PK) sampling, and efficacy evaluations.

Starting with the sentinel dose, one sentinel patient will be enrolled in the low-dose group and observed for up to 28 days. If no dose-limiting toxicity (DLT) occurs in the sentinel patient, enrollment will proceed to the medium-dose group. Initially, one patient will be enrolled in this group. If no DLT is observed, two additional patients will be enrolled in the medium-dose group. If no DLT occurs in any of these patients, escalation to the high-dose group will begin. If one DLT occurs, one additional patient will be enrolled in the same dose group; if ≥2 DLTs occur, the previous dose will be determined as the MTD.

The high-dose group will enroll three patients, with the possibility of expanding to six if needed. To ensure the trial can escalate to the anticipated effective dose, if no DLTs are observed in the low-, medium-, or high-dose groups, and no changes are observed in objective response rate or liver function indicators, the dose may be adjusted to 9 mg/kg. One patient will be enrolled at this dose level; if no DLT occurs, two additional patients will be enrolled.

If disease progression is observed at the 6-week efficacy assessment, subsequent treatment will involve CREPT-618 administration every two weeks in combination with pembrolizumab. Based on a comprehensive evaluation of safety and pharmacodynamic (PD) data from existing patients, the investigator may adjust the dosing frequency. If higher doses are tolerated and potential benefits are anticipated, dose escalation to a higher dose group is permitted within the same subject (allowed only once).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old.
* Diagnosis: Patients with histologically confirmed locally or advanced hepatocellular carcinoma (HCC) (BCLC stage C or ineligible for curative treatment).
* Hepatitis B Status: Inactive hepatitis B virus infection with negative HBV-DNA viral load.
* Informed Consent: Ability to understand and voluntarily sign the informed consent form.
* Prior Treatment: Failed prior standard treatment.
* ECOG Performance Status: ECOG performance status score of 0-2.
* Measurable Disease: Presence of at least one measurable lesion according to RECIST 1.1 criteria.
* Biomarker Status: Must be able to provide at least six unstained slides for testing, confirming both CREPT and ASGPR receptor positivity in liver cancer tissue. Alternatively, a tumor biopsy can be performed to confirm CREPT and ASGPR double positivity. H-score must be greater than 50% with a staining intensity of 2+.
* Organ Function: Acceptable major organ function as defined by the following laboratory values: Platelets ≥ 70 × 10^9/L Neutrophils ≥ 1.5 × 10^9/L Hemoglobin ≥ 90 g/L Prothrombin time prolongation ≤ 6 seconds Renal function: Creatinine clearance (Ccr) > 50 ml/min (calculated using the Cockcroft-Gault formula).
* Life Expectancy: Expected life expectancy of at least 3 months.
* Contraception: Male and female patients of childbearing potential must agree to use effective contraception (hormonal, barrier, or abstinence) during the study and for at least 6 months after the last dose of the study drug. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment.
* Compliance: Patients must be compliant and willing to adhere to follow-up procedures.

Exclusion Criteria:

- Prior Treatment:

a) Received systemic anti-tumor therapy (chemotherapy, radiotherapy, biological therapy, cytokine therapy, immunotherapy) or participated in other therapeutic clinical studies within 4 weeks prior to the first dose of the study drug. This includes nitrosourea drugs or mitomycin C within 6 weeks prior to the first dose. Exceptions: i) Oral fluoropyrimidine drugs or small molecule targeted agents received more than 2 weeks or 5 half-lives before the first dose (whichever is longer, but not exceeding 28 days).

ii) Traditional Chinese medicine for anti-tumor treatment received more than 2 weeks prior to the first dose.

iii) Palliative bone-directed radiotherapy. b) Planned to undergo major surgery within 28 days before the start of the study treatment (diagnostic biopsies are permitted).

c) Received systemic immunostimulants within 4 weeks or 5 half-lives (whichever is longer) prior to enrollment.

d) Used systemic corticosteroids (prednisone > 10 mg/d or equivalent dose) or other immunosuppressive drugs within 14 days before the start of study treatment. Exceptions include topical, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids, or short-term use of corticosteroids for prophylactic purposes.

* Autoimmune Disease: Active autoimmune disease or a history of autoimmune disease within the past 2 years. Exceptions: vitiligo, Graves' disease, Hashimoto's disease, or psoriasis that did not require systemic treatment within the past 2 years.
* Severe Liver Decompensation: Presence of any of the following symptoms or abnormal indicators of severe liver function decompensation: Refractory ascites (unresponsive to diuretics or requiring frequent paracentesis); Hepatic encephalopathy ≥ Grade 2 (West Haven criteria); History of or current spontaneous bacterial peritonitis (SBP);Hepatorenal syndrome; History of esophagogastric variceal bleeding (within the last 3 months); Hepatic hydrothorax, hepatopulmonary syndrome, portal vein thrombosis (complete occlusion), or other severe liver-related complications;
* Laboratory Values: Total bilirubin > 3 mg/dL (51.3 μmol/L) Albumin < 2.8 g/dL (28 g/L) INR > 2.3 or prothrombin time prolongation > 6 seconds ALT or AST > 3 times the upper limit of normal (ALT > 120 U/L, AST > 105 U/L) Serum sodium < 130 mmol/L Serum creatinine > 1.5 mg/dL (133 μmol/L);
* Severe Infection/Comorbidities:

  1. Positive for HIV or a known history of AIDS.
  2. Positive for Hepatitis C virus (anti-HCV or HCV-RNA). (Patients with Hepatitis B may be included if they are receiving and willing to continue antiviral treatment according to local guidelines).
  3. Interstitial lung disease, obstructive lung disease, active bronchospasm, or oxygen saturation < 93% ("pulmonary insufficiency"), or any other active or severe pulmonary disease that may cause severe respiratory distress.
* Unresolved Toxicity: Unresolved toxicities from prior anti-cancer treatment that have not recovered to ≤ Grade 1. Exceptions may include toxicities judged by the investigator to not pose a safety risk (e.g., alopecia, Grade 2 peripheral neuropathy, or stable hypothyroidism on hormone replacement therapy).
* Comorbidities: Uncontrolled diabetes (fasting blood glucose > 200 mg/dL or 11.1 mmol/L), severe cardiovascular disease (e.g., myocardial infarction within the last 6 months, unstable angina, NYHA Class III-IV heart failure), etc.
* Brain Metastases: Patients with symptomatic active brain or meningeal metastases, primary central nervous system (CNS) tumors, or CNS metastases that have failed local treatment. Patients with asymptomatic or stable CNS metastases for at least 28 days without steroid use and confirmed as stable on a screening scan may be included.
* Other Malignancies: A history of other active malignancies within 5 years prior to enrollment, excluding basal cell or squamous cell skin cancer, cervical carcinoma in situ, papillary thyroid cancer, ductal carcinoma in situ of the breast, or other malignancies for which the patient has been disease-free for more than 5 years.
* Vaccination: Received live attenuated vaccines within 28 days prior to the first dose of the study drug. During the study, no vaccines other than inactivated vaccines (e.g., inactivated influenza vaccine) are permitted.
* Prior Immunotherapy: History of immunotherapy (including anti-CTLA-4/anti-PD-L1 or other agents) with any unresolved irAEs > Grade 1 prior to the first dose, or a history of irAEs ≥ Grade 3. Also, known allergy to any component of the CREPT-618 formulation.
* Other: Received liver transplant evaluation or planned liver transplant within 4 weeks prior to the first dose, or planned during the study.

Psychological/Compliance Issues: Patients with a mental disorder or poor compliance.

Substance Abuse: Known history of alcohol or drug abuse.

Pregnancy/Lactation: Pregnant or lactating female patients. Pregnancy is defined as a positive laboratory test for human chorionic gonadotropin (hCG) within 7 days before starting the study drug.

Investigator Discretion: Any other severe physical or mental illness or abnormal laboratory finding that the investigator believes makes the patient unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | From enrollment to the end of treatment at 12 weeks
  Safety: Incidence of adverse events (AEs) (graded according to CTCAE v5.0)， Dose-limiting toxicity (DLT) and maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | baseline and after treatment (0.5h, 1h, 2h, 4h, 8h, 24h for first dose, 1h for second dose(day15) and third dose(day 29))
  Pharmacokinetics (PK): Peak plasma concentration (Cmax) of CREPT-618 in plasma.
Pharmacokinetics (PK) | baseline and after treatment (0.5h, 1h, 2h, 4h, 8h, 24h for first dose, 1h for second dose(day15) and third dose(day 29))
  half-life (t1/2) of CREPT-618 in plasma.
Pharmacokinetics (PK) | baseline and after treatment (0.5h, 1h, 2h, 4h, 8h, 24h for first dose, 1h for second dose(day15) and third dose(day 29))
  area under the curve (AUC0-∞) of CREPT-618 in plasma.
Pharmacodynamics(PD) | baseline and 6 weeks after treatment
  Analysis of changes in CREPT protein expression after treatment using immunohistochemical staining of puncture liver tumor tissue.
Preliminary Efficacy | about 2 years
  Tumor objective response rate (ORR, RECIST 1.1, iRECIST)
Preliminary Efficacy | about 2 years
  disease control rate (DCR)
Preliminary Efficacy | about 2 years
  progression-free survival (PFS)
Preliminary Efficacy | at baseline and 15 days after treatment.
  Measure quality of life score by EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire)
preliminary efficacy | about 2 years
  changes in serum AFP levels
Preliminary Efficacy | Baseline and 15 days after first treatment
  Measure quality of life score by EORTC QLQ-HCC18 (EORTC Quality of Life Questionnaire - Hepatocellular Carcinoma 18 )

OTHER OUTCOMES:
Biomarker analysis | Baseline and 6 weeks after treatment
  Paired comparisons will be conducted between post-biopsy tissue and pre-treatment archival formalin-fixed paraffin-embedded (FFPE) tissue blocks from the same patient. RNA sequencing and multiplex immunofluorescence (mIF) histochemistry will be employed to analyze alterations in the CREPT-associated signaling network and mechanisms underlying the remodeling of the tumor immune microenvironment following treatment.
  Blood-based biomarkers associated with sensitivity to CREPT-618 will be identified, including multiplex cytokine profiling, peripheral blood immune cell subset analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No